CLINICAL TRIAL: NCT05105893
Title: Effect of Date Fruit Consumption in Later Pregnancy on Length of Gestation Labor and Delivery of Nulliparous Women
Brief Title: Effect of Date Fruit Consumption in Later Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Salma Nisar, Resident OBGYN, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13102021
Record Dates: First submitted 2021-10-13; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Labor Long
Keywords: Dates; labour; period of gestation; delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dates group (Other): The experimental group of women was given several dates orally and instructed to take seven a day and record their consumption until the beginning of the active phase of labor. Seven pieces of dates are about 80g of daily consumption
  Interventions: Other: Dates group
- No dates (Other): This group wasnt provided dates.
  Interventions: Other: Dates group

INTERVENTIONS:
Other: Dates group — Seven dates to be provided to patients

SUMMARY:
EFFECT OF DATE FRUIT CONSUMPTION IN LATER PREGNANCY ON LENGTH OF GESTATION LABOR AND DELIVERY OF NULLIPAROUS WOMEN

DETAILED DESCRIPTION:
This randomized, controlled study was conducted at the Gynecology and Obstetrics department of Pak Emirates Military Hospital for Six months duration from Jan 2021 to June 2021. Ethical consent for the study was taken from the Ethical Committee. All participants have signed the written consent. Healthy primigravida's at more than 37 weeks of gestation with no prenatal complications (low-risk pregnancies) or chronic diseases were invited to contribute in the analysis.

The criteria of exclusion included all primigravida and non-primigravida with prenatal problems. Prenatal complications included placenta praevia, rupture of membranes, multiple pregnancies, diabetes, hypertension and additional health problems, fetal abnormalities, fetal growth restriction or any contraindication to delivery by vagina.

The females who met the eligibility criteria were contacted and provided information related to the analysis. In the preliminary phase of contact with potential volunteers, the study was presented as a participant's usage of dates to expedite delivery. The randomization arrangement was performed by means of sealed envelopes numbered from 1 to 10, equally allocated by randomization to the date-consumers and the group of control. Therefore, they will be allocated to dates consumer or control group recipients.

ELIGIBILITY:
Inclusion Criteria:

* All primigravidas at 37 or more weeks gestation with low risk pregnancies

Exclusion Criteria:

* Any antenatal complications Preterm pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All pregnant females at 37 weeks gestation or more with no complications
Enrollment: 142 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of date fruit consumption in later pregnancy on length of gestation | 6 months
  Effect of Intake of dates in later pregnancy on the period of gestation in weeks
Effect of date fruit consumption in later pregnancy on labour and delivery | 6 months
  To know the effect of dates intake on onset of labour whether it enhances the spontaneous onset of labour, avoiding any induction of labour and the time of 1st and 2nd stage of labour (in hours)

CONTACTS AND LOCATIONS:
Overall Officials: Salma Nisar, Principal Investigator — Resident
Locations (1):
- PEMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No